CLINICAL TRIAL: NCT00070031
Title: A Phase II Study of Intravenous Edotecarin (PHA-782615) in Patients With Anthracycline- and Taxane-Refractory or Chemoresistant Metastatic Breast Cancer
Brief Title: Edotecarin in Treating Women With Locally Advanced or Metastatic Breast Cancer That Has Not Responded to Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000329917; MSKCC-03056; PHARMACIA-EDOABC-4439-001
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2009-12

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — edotecarin

INTERVENTIONS:
Drug: edotecarin

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as edotecarin use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well edotecarin works in treating women with locally advanced or metastatic breast cancer that has not responded to previous chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antitumor activity of edotecarin in women with anthracycline- and taxane-refractory or chemoresistant locally advanced or metastatic breast cancer.

Secondary

* Determine the time to tumor response and duration of response in patients treated with this drug.
* Determine the overall survival of patients treated with this drug.
* Determine the clinical benefit of this drug in these patients.
* Determine the safety and tolerability of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive edotecarin IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months until disease progression.

PROJECTED ACCRUAL: A total of 31-65 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed primary adenocarcinoma of the breast

  * Locally advanced or metastatic disease
* Not amenable to surgery or radiotherapy with curative intent
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR 10 mm by CT scan
  * Not previously irradiated
* Meets 1 of the following criteria:

  * Previously treated with anthracycline and concurrent or sequential taxane therapy

    * Refractory to the most recent taxane-based chemotherapy, defined as 1 of the following:

      * Progressive disease during therapy or within 4 months of the last dose with or without documented response for advanced disease
      * Progressive disease within 6 months of completing taxane-based chemotherapy as neoadjuvant therapy
  * Resistant to prior chemotherapy, as defined by progressive disease within 6 months of completing prior chemotherapy for advanced disease
* No known brain metastases or carcinomatous meningitis* NOTE: *Baseline CT scan or MRI of the brain required if there is clinical suspicion of CNS metastases
* No spinal cord compression
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN (5 times ULN if liver involvement secondary to tumor is present)
* Albumin at least 3.0 g/dL

Renal

* Creatinine no greater than 1.5 mg/dL

Cardiovascular

* LVEF at least 50% or ULN by echocardiogram or MUGA
* None of the following within the past 6 months:

  * Myocardial infarction
  * Severe or unstable angina
  * Symptomatic congestive heart failure
  * Cerebrovascular accident or transient ischemic attack
  * Deep vein thrombosis or other significant thromboembolic event
* No ongoing cardiac dysrhythmias grade 2 or greater
* No atrial fibrillation of any grade

Pulmonary

* No pulmonary embolism within the past 6 months

Gastrointestinal

* No active inflammatory bowel disease
* No partial or complete bowel obstruction
* No chronic diarrhea

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known HIV positivity
* No active infection
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No other severe acute or chronic medical or psychiatric condition or laboratory abnormality that would preclude study participation or confound study results

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent biological response modifiers
* No concurrent immunotherapy
* No concurrent sargramostim (GM-CSF)
* No other concurrent granulocyte colony-stimulating factors

Chemotherapy

* See Disease Characteristics
* Prior adjuvant chemotherapy allowed
* No prior topoisomerase I inhibitors
* No more than 2 prior chemotherapy regimens for advanced disease
* No prior high-dose chemotherapy that required hematopoietic stem cell rescue
* No other concurrent chemotherapy

Endocrine therapy

* Prior adjuvant hormonal therapy or hormonal therapy for advanced/metastatic disease allowed provided that therapy is discontinued before study entry
* No concurrent hormonal therapy

Radiotherapy

* See Disease Characteristics
* No prior radiotherapy to more than 25% of the bone marrow
* No concurrent radiotherapy during and for 5 days after study treatment

  * Palliative radiotherapy allowed provided no more than 20% of the bone marrow is involved

Surgery

* No coronary/peripheral artery bypass graft within the past 6 months

Other

* Recovered from prior therapy (except alopecia or neurotoxicity)
* At least 4 weeks since any other prior therapy
* More than 4 weeks since prior investigational agents
* No concurrent enrollment on another clinical trial
* No other concurrent approved or investigational anticancer treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-06; Primary Completion 2006-04 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D. Seidman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Clifford A. Hudis, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States